CLINICAL TRIAL: NCT03046160
Title: The Effect of Scapulothoracic Mobilization on Cervical Pain and Range of Motion in Patients With Neck Pain and Scapular Dyskinesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Abrar AlSadiq, Master Student, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-PGS-2015-03-219
Record Dates: First submitted 2017-01-24; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Neck Pain
Keywords: PPT; Scapula; Intervention; Manual therapy; mobilization
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Movement

ARMS (2):
- experimental group (Experimental): where treatment will involve conventional and Manual therapy (Mobilization with movement)+ tape (postural correction of scapular anterior tilt)
  1. The Manual therapy (Mobilization with movement)intervention was of grade III mobilizations with movement performed in sitting for 6-10 repetitions for 3 sets
  2. tape (postural correction of scapular anterior tilt)
  3. A program of 12 neck and scapular exercises.
  Interventions: Other: Manual therapy (Mobilization with movement); Other: neck and scapular exercises.; Other: corrective tape
- control group (Active Comparator): treatment will consist of the conventional approach+ tape (postural correction of scapular anterior tilt)
  1. tape (postural correction of scapular anterior tilt)
  2. A program of 12 neck and scapular exercises.
  Interventions: Other: neck and scapular exercises.; Other: corrective tape

INTERVENTIONS:
Other: Manual therapy (Mobilization with movement) — grade III mobilizations with movement, performed in sitting for 6-10 repetitions for 3 sets
  Other Names: MWM
  Arms: experimental group
Other: neck and scapular exercises. — A program of 12 neck and scapular exercises.
Other: corrective tape — elastic tape used to correct the anterior tilt of the scapula

SUMMARY:
Background: Dyskinesia has been referred to as a major manifestation of affected muscle performance and neuromuscular control of the scapular stabilizers. Alterations around the scapula with muscular imbalances could facilitate or emphasize dysfunction in its surrounding structures through compressive and shear stresses created by abnormal pull through attachments. No studies have investigated the effect of scapular mobilization with movement on neck mobility and pain. Objective: To quantify the effects of utilizing a scapular mobilization with movement on cervical pain and range of motion as compared to conventional treatment under the presence of scapular dyskinesia. Design: an experimental case-control study. Setting: Dammam Medical Complex. Methods: thirty-four patients with chronic non-specific neck pain. Participants will be allocated to one of two groups: experimental group where treatment will involve conventional and manual interventions or the control group where treatment will consist of the conventional approach only. The manual intervention will consist of a sustained corrective scapular glide during neck movement in all directions. Measurements will include: Visual Analog Scale, pressure pain threshold, neck range of motion, scapular rotation measure and Neck Disability Index. Statistical analysis: all will be done using SPSS version 22.0 for Mac. Means and standard deviations will be given as descriptive statistics. Paired t-test will be used to study the effects of scapulothoracic mobilization and exercises on neck range of motion and pain intensity. Independent t-test will be used to compare the effects of the two interventions on pain intensity Key words: Pressure pain threshold; Scapula; Intervention, Manual therapy, mobilization.

DETAILED DESCRIPTION:
Participants: Males and females aging between 25 and 50 years referred from orthopedic clinic with chronic neck pain were included in the study. Recruitment extends through the time period extending from April 2016- April 2017) by notices to orthopedics department with measures of inclusion and exclusion. Data is being collected at Dammam Medical Complex.

Sample: 34 participants with non-specific chronic neck pain (≥ 3 months)

Procedures:

Patients were screened for eligibility through inclusion and exclusion criteria. Consent forms were discussed thoroughly by the researcher to the patient and signed before the start of the study. Assessment will include the following: Detailed subjective information, and the data collection sheet demographic data (e.g., name, age, sex and side of scapular dyskinesia) (Appendix 5). Dyskinesia was identified using the Scapular Dyskinesis Test with 5 repetitions of active shoulder flexion and abduction, bilaterally, while holding a weight with either hand (1.4 kg for patients weighing less than 68.1 kg and 2.3 kg for patients weighing more than 68.1 kg). This test has good reliability and validity (McClure, Tate et al. 2009, Tate, McClure et al. 2009). Neck range of motion as well as active, passive and accessory movements were all assessed. Measurements were obtained three times. First time, at baseline from the patient interview and recorded on a data collection sheet and the second one was taken after completion of 3 sessions of treatment. The last measurement was taken at the end of all sessions.

Patients were assigned with random allocation to one of 2 groups using a computer-generated sequence of numbers by an independent therapist. The groups are: 1) Manual therapy (MWM) + tape (postural correction of scapular anterior tilt) and 2) Control (conventional treatment + tape (postural correction of scapular anterior tilt) groups. The manual therapy intervention was of grade III mobilizations with movement, performed by a certified Mulligan practitioner, in sitting for 6-10 repetitions for 3 sets. Home exercises including cervical retraction, scapular retraction, deep neck flexors strengthening and active range of motion exercises of neck in all directions were all done during the session and at home with 10 seconds hold for 10 repetitions for 5 times a day and were added in the same sequence in both groups. When the experimental group showed significantly improved results, some patients in the control group receive 2 extra sessions after all study measurements were obtained. Frequency of the sessions was carried out as 3 sessions/ week/ 30-60 minutes (Miller, Gross et al. 2010).

Manual Therapy Technique: The patient was sitting in a good relaxed posture with the therapist standing at the opposite side of the affected scapula. Reaching across the trunk, the palm of the left hand was over the clavicle with the right hand controlling the scapular glide. Both hands applied corrective gliding force (grade III) to reposition the scapula to the optimal position using an adduction force along with posterior and external rotations of the scapula. While maintaining this position, the subject was asked to move his neck through the restricted movement point of pain onset and return to starting point. When the technique was indicated, the patient was able to achieve a considerably greater range without pain. When needed, further modifications of the humeral head repositioning could be introduced. MWM were repeated 6-10 times before reassessing the movement independent of scapular repositioning. If the pain improved, further 3 sets of 6-10 repetitions were carried out.

Taping technique to correct anterior scapular tilt: A water-resistant active, elastic and adhesive kinesiotape was used I this study. An I-shaped elastic tape was applied over the muscle belly of the upper Trapezius (UT). The tape started with its anchor fixed anteriorly at the coracoid process and travelled posteriorly over the belly of upper Trapezius fibers and along the course of its lower fibers to get its final anchor at the thoracic spine.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 25- 50 years.
2. A history of neck pain lasting 3 months or more prior to study start.
3. A score of greater than or equal to 5/50 on the Neck Disability Index (NDI)(Vernon 2008, Vernon 2008)
4. Presence of scapular dyskinesia.

Exclusion Criteria:

1. Previous cervical spine or shoulder surgery
2. Cervical radiculopathy (compressed cervical nerve root on its way out of the spine, mainly could be manifested by pain, weakness, and sensory deficits (Corey and Comeau 2014)
3. Presence of a severe systemic disease (as fibromyalgia, Chronic fatigue syndrome, Diabetes mellitus, Hypertension, Grave's disease, Systemic lupus erythematous, Rheumatoid arthritis, Sickle cell disease) or any other widespread musculoskeletal pain syndromes.
4. Participation in an exercise program for the neck or scapular muscles in the 6 months preceding the study.
5. Consumption of stimulants (caffeine and nicotine) or analgesic drugs for at least 8 hours before the study.
6. Manual therapy contraindications (e.g., inflammatory joint disease, spinal cord pathology, infections, severe osteoporosis, cancer).
7. Whiplash injury/fracture.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Neck pain ( centimeters on visual analog scale) | up to 12 months

SECONDARY OUTCOMES:
Scapular rotatory range of motion (degrees) | up to 12 months
neck disability index (percentage) | up to 12 months
neck range of motion (degrees) | up to 12 months
pressure pain threshold (k pascal) | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dammam Medical Complex, Dammam, Eastern Province, Saudi Arabia